CLINICAL TRIAL: NCT05445492
Title: Clinical Validation Study for Noninvasive Cardiopulmonary Management Device
Brief Title: Respiration Validation for CPM Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Analog Device, Inc. (Other)
Collaborators: Clayton Sleep Insititute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Resp CPM Validation Clayton
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Cardiopulmonary Disease
MeSH Terms: conditions — Pulmonary Heart Disease

STUDY DESIGN:
Intervention Model Description: Non-randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Healthy Cohort (Experimental): The target population for this cohort is healthy adult volunteers who do not have preexisting heart or lung conditions or illness. The goal is to recruit a participant population with a range of body types and BMIs and an approximately even split of genders and compare the reference device measurements to the test device.
  Interventions: Device: CPM Device

INTERVENTIONS:
Device: CPM Device — The CPM device and reference device are used simultaneous to validate the CPM device.

SUMMARY:
This study is designed to be a clinical validation study to ready the CPM System for FDA 510(k) submission. This study will be conducted as a prospective non-randomized. The study is non-significant risk since the CPM Device is noninterventional and noninvasive. The study is primarily designed to validate the accuracy of the respiration rate and the changes in relative tidal volume. All participants will be fitted with both the CPM Device as well as reference devices (capnography and ECG). Participants will be randomized between 4 procedures (A-D) which will determine the order of 10 exercises. Each exercise has about 2 minutes of device recording and two minutes of rest. Each exercise contains two positions: sitting up for one minute and lying down for one minute. For some exercises, the participant will be instructed to breathe at a certain rate (assisted by a metronome). For other exercises, the participants will breathe at a normal rate but change how deep the are breathing. For the last, all capnography reference devices will be removed, and an ECG reference device will be placed. After exercise 18, the participant will have all devices removed and the study visit will terminate. The participant will receive a safety follow-up call about 1 week after their visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 and who are willing and able to give informed consent
* Willing and able to participate in all activities related to this study, including trimming chest hair and wearing a reference device and the CPM wearable device
* Volunteers of any race, any gender
* Range of physiques
* Healthy

Exclusion Criteria:

* Injury or skin disturbance in the area of the test device
* Allergies or sensitivities to silicone/acrylic-based adhesive
* Pregnant
* Currently smokes cigarettes
* Has known respiratory conditions that might prevent them from following the study procedure such as:

  * Flu
  * Pneumonia/bronchitis
  * Shortness of breath/respiratory distress
  * Respiratory or lung surgery
  * Emphysema, COPD, lung disease
* Has self-reported heart or cardiovascular conditions such as chest pain, AFib, CHF, cardiomyopathy, or other conditions that could interfere with cardiopulmonary function
* Has other self-reported health conditions that could interfere with the breathing patterns and exercises detailed in the protocol (including wearing a capnography mask)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clayton Sleep Institute, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Cohort
Started | 41
Completed | 40
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Cohort
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (13.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 171.8 (11.5)
Height [Mean (Standard Deviation); unit: centimeters] | 171.8 (11.5)
Weight [Mean (Standard Deviation); unit: kilograms] | 82.7 (23.2)

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of CPM System Calculated RR Versus Reference Device Via Percent of Error Accuracy of Respiration Rate
Description: Percentage of respiration rate error within ± 2bpm. Acceptance criteria for clinical utility is >= 85%. The percentage of respiration rate within ± 2brpm was calculated by data points, regardless of its rate and breathing condition, which the CPM System did not screen, therefore reporting the numeric values. Each data point will produce binary result (True or False) if the error is within ± 2 brpm. Assuming this binary result follows a binominal distribution, its confidence interval is also calculated.
Time Frame: 90 minutes
Measure: Number (95% Confidence Interval); unit: Percent
Units Other Than Participants: device measurements
Groups:
- Supine Position: This arm includes measurement data from position 1 of a CPM System reading (supine position).
- Upright Position: This arm includes measurement data from position 2 of a CPM System reading (upright position).
Arm/Group | Supine Position | Upright Position
Number analyzed (Participants) | 40 | 40
Number analyzed (device measurements) | 360 | 360
Percent | 99.1 [97.4 to 99.8] | 98.5 [96.5 to 99.5]

2. Primary Outcome: Root Mean Squared Error (RMSE) of Respiration Rates From the CPM System vs Reference Device for Metronome Guided Breathing and Non-metronome Guided Breathing.
Description: First, the subject-specific linear fitting is performed after taking the natural log of both CPM's rTV and reference TV. Then, the residual errors in rTV after the fitting were calculated. Finally, all subject's residual errors are pooled together to calculate the root mean squared (RMS) residual relative errors. The confidence interval was calculated assuming the square of this error follows Chi-square distribution. This error characterized in a log-log domain is converted back to characterize a relative accuracy by taking an exponential of natural constant followed by subtraction of one. The RMS of residual error in % is characterized in this way because the linear fitting in the log-log domain and its residual errors represents faithful relative residual error regardless of an absolute value of TV.
Time Frame: 90 minutes
Measure: Number; unit: breath rates per minute (BRPM)
Units Other Than Participants: Device measurements
Arm/Group | Supine Position | Upright Position
Number analyzed (Participants) | 40 | 40
Number analyzed (Device measurements) | 360 | 360
breath rates per minute (BRPM)
  Root mean squared error for metronome guided breathing | 0.83 | 1.41
  Root mean squared error for non-metronome guided breathing | 1.03 | 0.97

3. Secondary Outcome: Performance of CPM System's ECG by % of CPM ECG Strip Equivalent to Lead II Strip
Description: Performance of CPM System's ECG is measurement by comparing CPM System ECG metrics to the reference device Lead II ECG strip. Clinicians reviewed the criteria below and decided if the CPM strip had equivalence to the Lead II strip.
Time Frame: device measurement (3 minutes)
Population: For 29 participants, a CPM lead strip and a Lead II ECG strip was generated.
Measure: Number; unit: % of CPM Strips Equivalent to Lead II
Units Other Than Participants: ECG Strips
Arm/Group | Healthy Cohort
Number analyzed (Participants) | 29
Number analyzed (ECG Strips) | 58
% of CPM Strips Equivalent to Lead II
  Quality QRS Presentation | 100
  QRS width measurability | 100
  Accurate Determination of QRS widening | 94
  QT interval measurability | 100
  A-Fib Rhythm Readability | 100

4. Secondary Outcome: ECG Accuracy Confirmation Comparing CPM Systems Generated ECG Metrics and Reference Lead II Generated ECG Metrics
Description: Determine the accuracy of CPM System's ECG metrics to the reference device. Results are displayed as mean error with standard deviation of error.
Time Frame: device measurement (3 minutes)
Population: For 29 participants, one ECG strip for CPM and one ECG strop for Lead II reference device were generated and compared.
Measure: Mean (Standard Error); unit: milliseconds (ms)
Units Other Than Participants: ECG Strips
Arm/Group | Healthy Cohort
Number analyzed (Participants) | 29
Number analyzed (ECG Strips) | 58
milliseconds (ms)
  Heart Rate (Beats per minute) | -0.2 (2.0)
  QRS witdh | 18.9 (10.8)
  QRS width (ms) excluding 8% of outliers | 17.4 (9.6)
  QT interval (ms) | 27.5 (40.9)
  QT interval (ms) excluding 8% of outliers | 20.3 (33.1)
  QTc interval | 27 (37.6)
  QTc interval excluding 8% f outliers | 20.4 (30.7)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Healthy Cohort
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT05445492/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT05445492/SAP_002.pdf